CLINICAL TRIAL: NCT05299749
Title: Real-time fMRI Neurofeedback as a Tool to Mitigate Auditory Hallucinations in Patients With Schizophrenia - R33 Phase
Brief Title: Real-time fMRI Neurofeedback in Patients With Schizophrenia and Auditory Hallucinations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston VA Research Institute, Inc. (Other)
Collaborators: Mclean Hospital (Other); Northeastern University (Other); Cambridge Health Alliance (Other)
Responsible Party: Principal Investigator, Margaret Niznikiewicz, Professor in Psychiatry, Boston VA Research Institute, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4R33MH113751-03 (NIH)
Record Dates: First submitted 2022-03-08; First posted 2022-03-29 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia; Auditory Hallucination; Treatment-resistant Schizophrenia
Keywords: Auditory-Hallucination; Connectivity; brain-activity; default-mode-network; superior temporal gyrus; Neurofeedback; MRI
MeSH Terms: conditions — Schizophrenia; Hallucinations; Schizophrenia, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- stg-rt-fMRI (Experimental): will receive feedback from the STG
  Interventions: Other: stg-rt-fMRI-Neurofeeback
- sham-rt-fMRI (Sham Comparator): will receive feedback from the motor cortex
  Interventions: Other: sham-rt-fMRI-Neurofeedback

INTERVENTIONS:
Other: stg-rt-fMRI-Neurofeeback — the patients will receive real-time feedback from the brain activity of the superior temporal gyrus
  Arms: stg-rt-fMRI
Other: sham-rt-fMRI-Neurofeedback — the patients will receive real-time feedback from the brain activity of the somato-motor cortex
  Arms: sham-rt-fMRI

SUMMARY:
Neurofeedback intervention aimed to regulate the superior temporal gyrus (STG) activation and default mode network (DMN) connectivity as well as to reduce the auditory hallucinations (AH) schizophrenia patients with medication resistant AH.

DETAILED DESCRIPTION:
Here, the investigators propose that neurofeedback aimed to regulate the superior temporal gyrus (STG) activation will not only lead to activation changes in the STG, but also to changes in the default mode network (DMN), as well as to reductions in AH, and that the brain and clinical changes will be correlated. The theoretical framework for the current proposal is an AH model that assumes that AH result from abnormalities in a network of regions including STG, and medial prefrontal cortex (MPFC) and posterior cingulate cortex (PCC), the two latter regions are core medial hubs of DMN that are related to self-referential processing. This model is supported by several theoretical papers and experimental evidence well as preliminary data by the investigators (PD). In both R61 and R33 the investigators will study SZ patients with medication resistant AH in the rt-fMRI intervention arm and in the sham-rt-fMRI arm. In both arms, the task and the rt-fMRI session structure will be identical. The SZ-intervention group will receive feedback from the STG while SZ-sham group will receive feedback from the motor cortex. In addition, 2 functional fMRI tasks will examine the effect of rt-fMRI neurofeedback and of sham-rt-fMRI on brain response. This R33 phase will consist of an SZ-intervention group (random n=52) that will receive 5 sessions of rt-fMRI feedback targeting STG, while SZ-sham group (random n=52) will receive 5 sham-rt-fMRI sessions. Based on our R61 phase data, the investigators predict that rt-fMRI feedback aimed at STG will reduce AH which will be, in turn, associated with reductions in the STG activation and in the DMN connectivity (i.e., brain changes achieved in R61 and replicated in R33) in SZ- intervention group only. Five sessions of rt-fMRI feedback will address the question of dose response at brain and clinical levels. The impact of rt-fMRI neurofeedback and of sham-rt-fMRI on AH (primary outcome), and on delusions, negative symptoms and working memory (WM) (exploratory outcome) will be assessed with clinical and neuropsychological measures. In an exploratory aim, based on the existing literature, the investigators predict the improvement in delusions, negative symptoms and in WM score, only post-rt-fMRI neurofeedback targeting the STG and not post-sham-rt-fMRI.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with SZ or schizoaffective disorder using DSM-5 criteria
* auditory hallucinations not responsive to pharmacology as determined by chart review and a clinical interview of SCID.

Exclusion Criteria:

* neurologic illness
* major head trauma
* electroconvulsive therapy
* alcohol or drug dependence
* alcohol or drug abuse within the past five years
* verbal IQ below 70

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
percent change in the STG BOLD signal, post- relative to pre-NFB | 0-4 weeks post intervention
  does real-time fMRI neurofidback reduce BOLD activity in STG, post NFB

SECONDARY OUTCOMES:
reduction in scores on Psychotic Symptoms Rating Scale, post- relative to pre, NFB | 0-4 weeks post intervention
  does real-time fMRI neurofidback reduce auditory hallucinations, post NFB
percent change in the MPFC-PCC connectivity measure, post- relative to pre-NFB. | 0-4 weeks post intervention
  Does real time NFB reduce connectivity in MPFC-PCC, post NFB

CONTACTS AND LOCATIONS:
Overall Officials: margaret niznikiewicz, Principal Investigator — Boston VA Research Institute, Inc.
Locations (1):
- Boston VA Healthcare System, Brockton, Brockton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Clinical, Cognitive and Imaging data will be made publicly available
Supporting Information: Study Protocol, SAP
Time Frame: after results are published in peer reviewed journal; in perpetuity
Access Criteria: researchers as confirmed by NIMH